CLINICAL TRIAL: NCT06610968
Title: Effects of Acute Vitamin D Supplementation on Testosterone in Young, Healthy Females: A Pilot Study
Brief Title: Acute Vitamin D Supplementation on Testosterone in Females
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Todd Schroeder, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HS-24-00403
Record Dates: First submitted 2024-09-17; First posted 2024-09-24 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Female Hormone Profile
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either a treatment or control group upon enrollment and blinded to group assignment. The treatment intervention will consist of three weeks of one 5000 IU cholecalciferol capsule (Pure Encapsulations, LLC) daily, with breakfast. The control group will also take a daily, with breakfast, placebo capsule (Zeebo) for the three-week intervention.
Who Masked: Participant
Masking Description: Single blinded intervention. Those measuring the blood samples' hormonal will also be blinded to the intervention group but will not have a role in data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D Group (Experimental): The treatment intervention will consist of three weeks of one 5000 IU cholecalciferol capsule (Pure Encapsulations, LLC) daily, with breakfast.
  Interventions: Dietary Supplement: Vitamin D (Cholecalciferol )
- Placebo Group (Placebo Comparator): The control group will also take a daily, with breakfast, placebo capsule (Zeebo) for the three-week intervention.
  Interventions: Dietary Supplement: Placebo Group

INTERVENTIONS:
Dietary Supplement: Vitamin D (Cholecalciferol ) — 5000 IU Vitamin D (as cholecalciferol) capsules (Vitamin D3 125 mcg [5,000 IU], Pure Encapsulation, LLC) daily
  Other Names: 5000 IU Vitamin D daily
  Arms: Vitamin D Group
Dietary Supplement: Placebo Group — One placebo capsule (Zeebo Imagine, Zeebo) daily.
  Other Names: Placebo (Zeebo) pill daily
  Arms: Placebo Group

SUMMARY:
Participation will take place over two visits to the Clinical Exercise Research Center (CERC) at the University of Southern California Health Sciences Campus.

On the first visit, height, weight, and body composition by bioelectrical impedance are recorded. Questionnaires and withdrawal of a sample of blood (1 tablespoon) are also completed. The intervention begins the day following the first visit. The intervention protocol consists of three weeks of consuming either a placebo capsule or a 5000 IU Vitamin D capsule daily and completing a daily survey.

The second visit to CERC immediately follows the 3-weeks intervention. In this visit, the same blood sampling protocol will be completed. The assignment of the intervention will be randomized (i.e., rolling a die), and participants are blinded to group assignment.

DETAILED DESCRIPTION:
High-dose Vitamin D supplementation significantly increases testosterone in men, but research about Vitamin D's effect on testosterone in young, healthy females is limited [1]. However, testosterone is a critical hormone for many physiologic functions in females including maintenance of reproductive health, cognitive function, body composition, mental health, bone density, muscle strength, and much more. Thus, this study aims to investigate the effect of Vitamin D supplementation on testosterone and gonadotropin concentrations in premenopausal, healthy females. The study investigators hypothesize that Vitamin D supplementation will result in a significant increase in circulating Vitamin D [25(OH)D], testosterone, and sex hormone modulators (i.e., gonadotropins and SHBG) concentrations in pre-menopausal females and that the magnitude of testosterone increase will be inversely related to fat mass and BMI. 20 young, healthy females will be randomized to either a treatment or placebo group for a three-week intervention, where the control group will take 5000 IU of Vitamin D orally, daily and the placebo group will take a placebo capsule orally, daily. Circulating Vitamin D, testosterone, gonadotropin, and SHBG concentrations will be assessed via serum pre- and post-intervention. Two-tailed unpaired t-test will be conducted to assess the relative change in total testosterone and free testosterone levels between the groups. Additionally, correlation analyses will be performed for correlations between body composition metrics and 25(OH)D, testosterone, and sex hormone modulator concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Assigned female at birth
* 18 to 35 years of age
* No chronic diseases affecting the uptake of Vitamin D or causing Vitamin D sensitivity (e.g., sarcoidosis, tuberculosis, Wegener's granulomatosis, other forms of vasculitis, inflammatory bowel diseases, etc.) [21]
* Completion and signature of the informed consent document
* Non-pregnant or trying to become pregnant
* No supplementation with Vitamin D within three months of enrollment
* No documented gynecological disease (e.g., PCOS, endometriosis, etc.)
* Weight greater than or equal to 110 lbs

Exclusion Criteria:

* Pregnant
* Supplementation with Vitamin D within three months of enrollment
* Taking exogenous hormones
* Documented gynecological disease (e.g., PCOS, endometriosis, etc.)
* Suffering from chronic diseases affecting the uptake of Vitamin D or causing Vitamin D sensitivity (e.g., sarcoidosis, tuberculosis, Wegener's granulomatosis, other forms of vasculitis, inflammatory bowel diseases, etc.) [21]
* Weight less than 110 lbs

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Hormonal Effects of Vitamin D in Young, Healthy Women | 3 weeks
  The primary objective is to evaluate the effect of acute Vitamin D supplementation on systemic Vitamin D, testosterone, and sex hormone modulators in pre-menopausal, healthy females. Circulating testosterone (total testosterone and free testosterone) concentrations (ng/dL) will be assessed via serum pre- and post-Vitamin D intervention.
Hormonal Effects of Vitamin D in Young, Healthy Women | 3 weeks
  The primary objective is to evaluate the effect of acute Vitamin D supplementation on systemic Vitamin D, testosterone, and sex hormone modulators in pre-menopausal, healthy females. Circulating Vitamin D [25(OH)D] concentrations (ng/dL) will be assessed via serum pre- and post-Vitamin D intervention.
Hormonal Effects of Vitamin D in Young, Healthy Women | 3 weeks
  The primary objective is to evaluate the effect of acute Vitamin D supplementation on systemic Vitamin D, testosterone, and sex hormone modulators in pre-menopausal, healthy females. Circulating gonadotropins (LH and FSH) concentrations (IU/L) will be assessed via serum pre- and post-Vitamin D intervention.
Hormonal Effects of Vitamin D in Young, Healthy Women | 3 weeks
  The primary objective is to evaluate the effect of acute Vitamin D supplementation on systemic Vitamin D, testosterone, and sex hormone modulators in pre-menopausal, healthy females. Circulating SHBG concentrations (nmol/L) will be assessed via serum pre- and post-Vitamin D intervention.

SECONDARY OUTCOMES:
Effects of Body Composition on Hormonal Changes Due to Vitamin D Supplementation in Young, Healthy Women | 3 weeks
  Secondary analyses will evaluate the effect of body composition on change in testosterone concentration due to acute Vitamin D supplementation of pre-menopausal, healthy females. Testosterone (TT and FT) concentrations will be correlated with body composition metrics, i.e. fat and fat-free mass (kg), pre- and post-Vitamin D intervention.
Effects of Body Composition on Hormonal Changes Due to Vitamin D Supplementation in Young, Healthy Women | 3 weeks
  Secondary analyses will evaluate the effect of body composition on change in testosterone concentration due to acute Vitamin D supplementation of pre-menopausal, healthy females. Testosterone (TT and FT) concentrations will be correlated with body composition metrics, i.e. BMI (kg/m^2) as measured from height (m) and weight (kg), pre- and post-Vitamin D intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Giuliet L Kibler, Principal Investigator — University of Southern California - Division of Biokinesiology and Physical Therapy
Locations (1):
- University of Southern California Health Sciences Campus Center for Health Professions, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pilz S, Frisch S, Koertke H, Kuhn J, Dreier J, Obermayer-Pietsch B, Wehr E, Zittermann A. Effect of vitamin D supplementation on testosterone levels in men. Horm Metab Res. 2011 Mar;43(3):223-5. doi: 10.1055/s-0030-1269854. Epub 2010 Dec 10. PMID 21154195